CLINICAL TRIAL: NCT03796182
Title: A PHASE 1, RANDOMIZED, 2-WAY CROSSOVER, OPEN LABEL STUDY TO ESTIMATE THE EFFECT OF PF-04965842 ON MATE1/2K ACTIVITY, USING METFORMIN AS A PROBE, IN HEALTHY PARTICIPANTS
Brief Title: Study of PF 04965842 Effect on MATE1/2K Activity in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B7451034; DDI (Other: Alias Study Number); 2018-003683-31 (EudraCT Number)
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Healthy
Keywords: Phase 1; Metformin; Atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Metformin; abrocitinib

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, randomized, 2 way crossover, open label study of the effect of PF 04965842 on metformin PK in healthy adult participants. The effect of PF 04965842 on N1 methylnicotinamide (NMN) PK and its correlation to the effect on metformin PK will also be assessed.
  A total of approximately 12 healthy male and/or female participants will be enrolled in the study so that approximately 6 participants will be enrolled in each treatment sequence. Each treatment sequence will consist of 2 periods. Participants who discontinue from the study may be replaced at the sponsor's discretion. The replacement participant will receive the same treatment sequence as the participant who discontinued.
  Participants will be screened within 28 days of the first dose of investigational product. Participants will report to the clinical research unit (CRU) the day prior to Day 1 (ie Day -1) dosing in Period 1 for both treatment sequences. In both sequences, participants will remain in the CRU for
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): Patients in sequence 1 will received treatment A (metformin) in Period 1 then complete at least 4 days of washout and continue to period 2 where treatment B (PF-04965842 + metformin) will be administered.
  Interventions: Drug: Metformin; Drug: PF-04965842
- Sequence 2 (Experimental): Patients in Sequence 2 will start treatment B (PF-04965842 + metformin) then go through a washout period of at least 4 days and continue to Period 2 where treatment A (metformin) will be administered.
  Interventions: Drug: Metformin; Drug: PF-04965842

INTERVENTIONS:
Drug: Metformin — Commercially available metformin (GLUCOPHAGE®) as 500 mg tablets.
  Other Names: Glucophage
Drug: PF-04965842 — PF 04965842 100 mg tablets

SUMMARY:
This is a Phase 1, randomized, 2 way crossover, open label study of the effect of PF-04965842 on metformin (a probe for MATE1/2K activity) PK in healthy adult participants. The effect of PF-04965842 on N1-methylnicotinamide (NMN; an endogenous biomarker for MATE1/2K) PK and its correlation to the effect on metformin PK will also be assessed. Participants will be randomized to 1 of 2 treatment sequences as described below. A total of 12 healthy male and/or female participants will be enrolled in the study so that 6 participants will be enrolled in each treatment sequence. Each treatment sequence will consist of 2 periods.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, 2 way crossover, open label study of the effect of PF-04965842 on metformin (a probe for MATE1/2K activity) PK in healthy adult participants. The effect of PF-04965842 on N1-methylnicotinamide (NMN; an endogenous biomarker for MATE1/2K) PK and its correlation to the effect on metformin PK will also be assessed. Participants will be randomized to 1 of 2 treatment sequences as described below. A total of 12 healthy male and/or female participants will be enrolled in the study so that 6 participants will be enrolled in each treatment sequence. Each treatment sequence will consist of 2 periods. Participants who discontinue from the study may be replaced at the sponsor's discretion. The replacement participant will receive the same treatment sequence as the participant who discontinued.

Participants will be screened within 28 days of the first dose of investigational product. Participants will report to the clinical research unit (CRU) the day prior to Day 1 (ie Day -1) dosing in Period 1 for both treatment sequences. In both sequences, participants will remain in the CRU for a total of 8 days and 7 nights (including Period 1 and Period 2). There will be a minimum 4 day washout period between metformin dosing events. NMN and metformin PK will be assessed in plasma and urine over 24 and 48 hours, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are overtly healthy as determined by medical evaluation including a detailed medical history, complete physical examination, laboratory tests, and cardiovascular tests.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Female participants who are of child bearing potential must not be intending to become pregnant, currently pregnant, or lactating.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Capable of giving signed informed consent.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* History of human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus infection; positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), or hepatitis C virus antibody (HCVAb).
* Other acute or chronic medical or psychiatric condition including recent (within the past year).
* Evidence or history of clinically significant dermatological condition (eg, atopic dermatitis or psoriasis) or visible rash present during physical examination.
* Clinically relevant history of lactic acidosis.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of investigational product.
* A positive urine drug test.
* Selected laboratory abnormalities.
* History of regular alcohol consumption exceeding 14 drinks/week for female participants or 21 drinks/week for male participants (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months before screening.
* Known relevant history of elevated liver function tests (LFTs).
* History of tuberculosis (TB) (active or latent)
* Any history of chronic infections, any history of recurrent infections, any history of latent infections, or any acute infection within 2 weeks of baseline.
* History of disseminated herpes zoster, or disseminated herpes simplex, or recurrent localized dermatomal herpes zoster.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Vourvahis M, Byon W, Chang C, Le V, Diehl A, Graham D, Tripathy S, Raha N, Luo L, Mathialagan S, Dowty M, Rodrigues AD, Malhotra B. Evaluation of the Effect of Abrocitinib on Drug Transporters by Integrated Use of Probe Drugs and Endogenous Biomarkers. Clin Pharmacol Ther. 2022 Sep;112(3):665-675. doi: 10.1002/cpt.2594. Epub 2022 May 9. PMID 35344588
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451034

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 12 healthy participants were enrolled in the study and 6 participants were assigned in each of the 2 treatment sequences, all receiving study treatment.
Groups:
- Metformin Then Metformin + PF-04965842: Participants were administered a single oral dose of metformin 500 mg on Day 1 in Period 1 followed by a washout period of at least 4 days. Then in Period 2 participants were administered a single oral dose of metformin 500 mg on Day 1 along with oral doses of PF-04965842 200 mg once daily (QD) for 2 days on Days 1-2.
- Metformin + PF-04965842 Then Metformin: Participants were administered a single oral dose of metformin 500 mg on Day 1 along with oral doses of PF-04965842 200 mg QD for 2 days on Days 1-2 in Period 1 followed by a washout period of at least 4 days. Then in Period 2 participants were administered a single oral dose of metformin 500 mg on Day 1.
Period: Period 1
Arm/Group | Metformin Then Metformin + PF-04965842 | Metformin + PF-04965842 Then Metformin
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | Metformin Then Metformin + PF-04965842 | Metformin + PF-04965842 Then Metformin
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Metformin Then Metformin + PF-04965842 | Metformin + PF-04965842 Then Metformin
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All 12 participants who were randomized to study treatment.
Groups:
- All Participants: This reporting group refers to the total 12 participants who were enrolled in the study.
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.0 (8.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Renal Clearance (CLr) of Metformin
Description: CLr was calculated as cumulative amount of drug recovered unchanged in urine during the dosing interval (Ae) divided by area under the plasma concentration time-curve from time zero to end of dosing interval (AUCtau).
Time Frame: For both Period 1 and Period 2 at intervals of 0-12, 12-24, 24-36, and 36-48 hours post metformin dose
Population: This analysis population was defined as all participants randomized and treated who had at least 1 of the PK parameters of primary interest in at least 1 treatment period. Overall number of participants analyzed referred to participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: litre per hour (L/hr)
Groups:
- Metformin + PF-04965842: This reporting group refers to the participants who were randomized to the group of concomitantly single oral administration of metformin 500 mg QD on Day 1 and oral administration of PF-04965842 200 mg QD for 2 days on Days 1-2 in either of the periods.
- Metformin: This reporting group refers to the participants who were randomized to the group of single oral administration of metformin 500 mg QD on Day 1 in either of the periods.
Arm/Group | Metformin + PF-04965842 | Metformin
Number analyzed (Participants) | 11 | 12
litre per hour (L/hr) | 32.18 (39) | 33.33 (28)
Statistical Analysis 1: Comparison: Metformin + PF-04965842 vs Metformin; Test type: Equivalence — The corresponding 90% confidence intervals equivalence criteria was (80%, 125%) acceptance range; Ratio = 98.50, 90% CI 2-sided [82.09 to 118.20]

2. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) of Metformin
Description: AUCinf is a measure of the serum concentration of the drug over time. It was used to characterize drug absorption.
Time Frame: Pre-dose and at 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose of metformin on Day 1 for both Period 1 and Period 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Metformin + PF-04965842 | Metformin
Number analyzed (Participants) | 8 | 11
nanogram*hour per milliliter (ng*hr/mL) | 5050 (16) | 5202 (19)
Statistical Analysis 1: Comparison: Metformin + PF-04965842 vs Metformin; Test type: Equivalence — The corresponding 90% confidence intervals equivalence criteria was (80%, 125%) acceptance range; Ratio = 93.49, 90% CI 2-sided [85.15 to 102.65]

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Metformin
Description: Cmax is maximum observed plasma concentration.
Time Frame: as for outcome 2
Population: This analysis population was defined as all participants randomized and treated who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Metformin + PF-04965842 | Metformin
Number analyzed (Participants) | 12 | 12
nanogram per milliliter (ng/mL) | 634.7 (14) | 720.7 (20)
Statistical Analysis 1: Comparison: Metformin + PF-04965842 vs Metformin; Test type: Equivalence — The corresponding 90% confidence intervals equivalence criteria was (80%, 125%) acceptance range; Ratio = 88.07, 90% CI 2-sided [80.99 to 95.76]

4. Secondary Outcome: Time for Cmax (Tmax) of Metformin
Description: Tmax of metformin administrated with or without PF-04965842.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours (hrs)
Arm/Group | Metformin + PF-04965842 | Metformin
Number analyzed (Participants) | 12 | 12
Hours (hrs) | 4.00 [2.00 to 4.00] | 4.00 [1.00 to 4.00]

5. Secondary Outcome: Area Under the Plasma Concentration Time Profile From Time 0 to the Time of Last Quantifiable Concentration (AUClast) of Metformin
Description: AUClast of metformin administrated with or without PF-04965842.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Metformin + PF-04965842 | Metformin
Number analyzed (Participants) | 12 | 12
ng*h/mL | 4849 (18) | 5145 (18)
Statistical Analysis 1: Comparison: Metformin + PF-04965842 vs Metformin; Test type: Equivalence — The corresponding 90% confidence intervals equivalence criteria was (80%, 125%) acceptance range; Ratio = 94.25, 90% CI 2-sided [88.19 to 100.73]

6. Secondary Outcome: Apparent Clearance (CL/F) of Metformin
Description: CL/F is a quantitative measure of the rate at which drug was removed from the blood.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Metformin + PF-04965842 | Metformin
Number analyzed (Participants) | 8 | 11
L/hr | 98.97 (16) | 96.13 (19)

7. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Metformin
Description: Vz/F is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)
Arm/Group | Metformin + PF-04965842 | Metformin
Number analyzed (Participants) | 8 | 11
liter (L) | 1087 (42) | 1211 (37)

8. Secondary Outcome: Terminal Half-life (t1/2) of Metformin
Description: t1/2 is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Metformin + PF-04965842 | Metformin
Number analyzed (Participants) | 8 | 11
hrs | 8.318 (4.2508) | 9.261 (3.5165)

9. Secondary Outcome: Cumulative Amount of Drug Recovered Unchanged in Urine From 0 to 48 Hours (Ae) of Metformin
Description: Ae is the cumulative amount of drug recovered unchanged in urine during the dosing interval. Cumulative amount was calculated as sum of urine drug concentration in sample volume for each collection interval. Sample volume = (urine weight in gram [g]/1.020), where 1.020 g/mL is the approximate specific gravity of urine.
Time Frame: For both Period 1 and Period 2 at intervals of 0-12, 12-24, 24-36, and 36-48 hours post metformin dose
Population: as for outcome 1
Measure: Median (Full Range); unit: milligram (mg)
Arm/Group | Metformin + PF-04965842 | Metformin
Number analyzed (Participants) | 11 | 12
milligram (mg) | 168.0 [70.7 to 210] | 170.5 [114 to 248]

10. Secondary Outcome: Percent of Dose Recovered Unchanged in Urine From 0 to 24 Hours (Ae%) of Metformin
Description: Ae% is percent of dose recovered unchanged in urine from 0 to 24 hours post-dose of metformin.
Time Frame: For both Period 1 and Period 2 at intervals of 0-12 and 12-24 hours post metformin dose
Population: as for outcome 1
Measure: Median (Full Range); unit: percentage of dose
Arm/Group | Metformin + PF-04965842 | Metformin
Number analyzed (Participants) | 11 | 12
percentage of dose | 33.60 [14.1 to 42.0] | 34.05 [22.7 to 49.7]

11. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Laboratory parameters included: hematology (hemoglobin, hematocrit, erythrocytes, ery. mean corpuscular volume, ery. mean corpuscular hemoglobin, ery. mean corpuscular HGB concentration, platelets, leukocytes, lymphocytes, neutrophils, basophils, eosinophils, monocytes, activated partial thromboplastin time, prothrombin time, prothrombin intl. normalized ratio, large unstained cells/leukocytes and large unstained cells), clinical chemistry (bilirubin, direct bilirubin, indirect bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, protein, albumin, blood urea nitrogen, urea, creatinine, urate, sodium, potassium, chloride, calcium, bicarbonate, urobilinogen and glucose -FASTING), urinalysis (specific gravity, pH, urine glucose, ketones, urine protein, urine hemoglobin, urine bilirubin, nitrite and leukocytes). Clinical significance of laboratory parameters is determined at the investigator's discretion.
Time Frame: Screening (within 28 days prior to Day 1) to Day 7
Population: This analysis population was defined as all participants randomly assigned to investigational product and who took at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin + PF-04965842 | Metformin
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

12. Secondary Outcome: Number of Participants With Categorical Vital Signs Meeting Pre-defined Criteria
Description: Criteria for change in vital signs: pulse rate value less than (<) 40 beats per minute (bpm) or value over than (>) 120 bpm, systolic blood pressure (SBP) value < 90 millimeter of mercury (mmHg) or change from baseline (Chg) equal to or over than (≥) 30 mmHg increase or ≥ Chg 30 mmHg decrease, diastolic blood pressure (DBP) value < 50 mmHg or Chg ≥ 20 mmHg increase or Chg ≥ 20 mmHg decrease.
Time Frame: Screening (within 28 days prior to Day 1) to Day 7
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin + PF-04965842 | Metformin
Number analyzed (Participants) | 12 | 12
Participants
  Supine DBP Value < 50 mmHg | 0 | 0
  Supine DBP Chg ≥ 20 mmHg increase | 0 | 0
  Supine DBP Chg ≥ 20 mmHg decrease | 0 | 0
  Supine pulse rate Value < 40 bpm | 0 | 0
  Supine pulse rate Value > 120 bpm | 0 | 0
  Supine SBP Value < 90 mmHg | 0 | 0
  Supine SBP Chg ≥ 30 mmHg increase | 0 | 0
  Supine SBP Chg ≥ 30 mmHg decrease | 0 | 0

13. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) (All Causalities and Treatment-related)
Description: AEs with all causalities were any untoward medical occurrences in a study subject administered a product or medical device which did not necessarily had causal relationship with the treatment or usage. An SAE was an AE resulting in any of the following endpoints or deemed significant for any other reason: death; life threatening (immediate risk of death); inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; or considered to be an important medical event. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment-emergent are events between first dose of study drug and up to 35 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Day 1 up to Day 40 (35 days after the last dose of metformin)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin + PF-04965842 | Metformin
Number analyzed (Participants) | 12 | 12
Participants
  AEs (all causalities) | 6 | 4
  AEs (treatment-related) | 5 | 4
  SAEs (all causalities) | 0 | 0
  SAEs (treatment-related) | 0 | 0

14. Secondary Outcome: Percentage of Participants With Treatment-Emergent AEs and SAEs (All Causalities and Treatment-related)
Description: as for outcome 13
Time Frame: Day 1 up to Day 40 (35 days after the last dose of metformin)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Metformin + PF-04965842 | Metformin
Number analyzed (Participants) | 12 | 12
percentage of participants
  AEs (all causalities) | 50.0 | 33.3
  AEs (treatment-related) | 41.7 | 33.3
  SAEs (all causalities) | 0.0 | 0.0
  SAEs (treatment-related) | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 40 (35 days after the last dose of metformin)
Arm/Group | Metformin + PF-04965842 | Metformin
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 6/12 | 4/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin + PF-04965842 (N=12) | Metformin (N=12)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT03796182/SAP_000.pdf
  • Study Protocol (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT03796182/Prot_001.pdf